CLINICAL TRIAL: NCT07367295
Title: Prospective Clinical Study, Using a Medical Device as an Adjuvant in the Treatment of Fungal (Candidiasis) and Bacterial Infections: Evaluation of the Safety and Efficacy of Rephegyn Vaginal Ovules
Brief Title: Prospective Clinical Study, Using a Medical Device (RepHegyn) as an Adjuvant in the Treatment of Fungal (Candidiasis) and Bacterial Infections
Status: Not yet recruiting | Type: Observational
Sponsor: Innate srl (Industry)
Responsible Party: Sponsor
Other Study IDs: MD 07b/2025/Rephe
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Bacterial Infections; Treatment of Fungal Infections, Candidiasis
Keywords: candidiasis; bacterial infection; RepHegyn; pH restoring; barrier action
MeSH Terms: conditions — Bacterial Infections; Candidiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Age between 18 and 75 years, female

SUMMARY:
The medical device It is indicated to promote the re-epithelialization processes of the vaginal mucosa, in the prevention of vaginal conditions of bacterial and fungal origin, and as an adjuvant in their treatment.

The primary efficacy endpoint is based on the VAS symptom score (abnormal vaginal discharge, lower abdominal pain, dysuria, burning micturition, dyspareunia, vulvar irritation, and itching on a 10-point scale), specifically the percentage of patients with therapeutic success, defined as resolution of signs and symptoms of recurrent bacterial and fungal infections (total symptom score <2) at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Signed written informed consent.
* At least two subjective symptoms and two objective signs (at least moderate) of vaginal inflammation due to infection. Vaginal inflammation will be assessed based on six subjective symptoms (burning, pain, itching, irritation, dyspareunia, and dysuria) and four objective signs (swelling, vaginal discharge typical of the infection, pH, and presence of abrasion/erosion).
* Confirmed recurrent bacterial vaginosis and candidiasis.
* Patient able to maintain a patient diary during the study.
* Patient is able to read and understand the language and content of the study materials, understands the requirements for follow-up visits, is willing to provide information at scheduled assessments, and is willing and able to comply with study requirements.

Exclusion Criteria:

* Patients who do not sign the informed consent form
* Other gynecological diseases, immunosuppressive diseases (e.g., HIV infection), or who are immunocompromised for reasons such as corticosteroid therapy, chemotherapy, anti-angiogenic agents, or immunosuppressants, patients with diabetes
* Patients receiving antibiotics, anti-inflammatory agents, analgesics, antineoplastic drugs, or immunosuppressants within 4 weeks prior to study inclusion
* History of connective tissue diseases, e.g., systemic lupus erythematosus, systemic sclerosis, Sjogren's syndrome, or mixed connective tissue disease
* Known allergy to any component of the device
* Subjects unable to understand the informed consent form or who have a high likelihood of non-compliance with study procedures and/or non-completion of the study according to the investigator's judgment
* Pregnancy and breastfeeding
* Time between the last day of the last menstrual period and the baseline visit >16 days or ≤5 days (for non-menopausal subjects).
* Participation in other clinical studies

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female: form 18 - 75 years old
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
efficacy endpoint: VAS score for symptoms | "From enrollment to the end of treatment at 12 days (evaluation after menstrual cycle)
  The primary efficacy endpoint is based on the VAS score for symptoms (abnormal vaginal discharge, lower abdominal pain, dysuria, burning micturition, dyspareunia, vulvar irritation, and itching on a 10-point scale), specifically the percentage of patients with therapeutic success, defined as resolution of signs and symptoms of recurrent bacterial and fungal infections (total symptom score <2) at the end of treatment reported below.

SECONDARY OUTCOMES:
efficacy: evaluation of pH | "From enrollment to the end of treatment at 12 days (after menstrual cycle)
  evaluation of pH with instrument for pH
efficacy: VAS evaluation | From enrollment to the end of treatment at 12 days (after menstrual cycle)
  The change from the semi-quantitative baseline score, expressed both for individual signs and symptoms and for their sum (total symptom VAS)
safety endpoint | From enrollment to the end of treatment at 12 days (after menstrual cycle)
  The safety and tolerability of the treatments will be evaluated by investigating local and expected adverse events, as a consequence of the application of the product and any other adverse events occurring during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Rhodense, Dipartimento di ginecologia e ostetricia, Viale Forlanini 95, Garbagnate Milanese, Michigan, Italy

IPD SHARING:
Plan to Share IPD: No